CLINICAL TRIAL: NCT02493790
Title: Impact of Cognitive Dysfunction in Chronic Obstructive Pulmonary Disease on Performance in Cognitive-motor Dual Task Situation
Brief Title: Cognitive Dysfunction in COPD Patients : Role in the Performance of Cognitive-motor Dual Task Situation?
Acronym: DysCo
Status: Completed | Type: Observational
Sponsor: 5 Santé (Other)
Collaborators: Groupe 5 Santé (Unknown)
Responsible Party: Sponsor
Other Study IDs: 5S-DYSCO
Record Dates: First submitted 2015-06-30; First posted 2015-07-10 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: cognitive dysfunction; Activity of Daily Living; interference; rehabilitation; cognitive-motor dual task
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Volunteers: Cognitive and motor performances were measured in a single and dual task situations.
  Interventions: Other: Cognitive and motor performances
- COPD patients: Cognitive and motor performances were measured in a single and dual task situations, before rehabilitation, and compared to those of healthy subjects. Then, Chronic Obstructive Pulmonary Disease patients were re-evaluated after rehabilitation.
  Interventions: Other: Cognitive and motor performances

INTERVENTIONS:
Other: Cognitive and motor performances

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a respiratory disease starting point characterized by multiple systemic effects as cognitive dysfunction. This one seems to have an impact in activity daily living, considered mainly as a cognitive-motor dual task situations. Yet to date, no study has specifically focused in the cognitive-motor performance in patients with COPD or on the effects during a rehabilitation program. The main objective of this work was to evaluate the impact of cognitive dysfunction in COPD, comparing performance between COPD patients and healthy subjects in a single and dual task cognitive-motor situation. The secondary objective was to assess the impact of a rehabilitation program on these performances.

ELIGIBILITY:
Inclusion Criteria:

* Male or female about 40 to 80 years old
* COPD patient (Tiffeneau <70%); stage moderate to severe (Stage 2,3 and 4) with or without oxygen therapy (>15h/day)
* Written and informed consent of the subject
* Authorization to physical activity referring doctor in the clinic
* Comorbidities no dominating

Exclusion Criteria:

* Subject with neurological pathology, cognitive or psychiatric
* Subject with pain and / or plantar injuries
* Subject has a prosthetic knee and / or hip.
* Subject requiring walking aid (cane, walker, etc.)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients, entered in a rehabilitation program in Clinique du Souffle were included
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Variability of Cognitive performances in a single and dual task situations | 3 months
  Cognitive performance were determined by error count and number of substraction during a counting task.
Variability of motor performances in a single and dual task situations | 3 months
  Motor performance were determined by variability of length and surface of postural condition and by step variability in locomotion condition

SECONDARY OUTCOMES:
Effect of rehabilitation program on Cognitive performances in a single and dual task | 3 months
  Comparison before and after rehabilitation program of counting task (number of substraction and error count)
Effect of rehabilitation program on motor performances in a single and dual task | 3 months
  Comparison before and after rehabilitation program of variability of length and surface of postural condition and step variability in locomotion condition